CLINICAL TRIAL: NCT00938717
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial of Linaclotide Administered Orally for 26 Weeks in Patients With Irritable Bowel Syndrome With Constipation
Brief Title: Trial of Linaclotide in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-302
Record Dates: First submitted 2009-07-12; First posted 2009-07-14 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: IBS
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Linaclotide or Matching Placebo
- 290 μg Linaclotide (Experimental)
  Interventions: Drug: Linaclotide or Matching Placebo

INTERVENTIONS:
Drug: Linaclotide or Matching Placebo — Linaclotide or Matching Placebo, administered orally, once daily, for the duration of the trial

SUMMARY:
The purpose of this study is to determine the safety and efficacy of linaclotide administered to patients with Irritable Bowel Syndrome with Constipation (IBS-C).

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a colonoscopy according to the AGA criteria, with no clinically significant findings
* Patient has successfully completed protocol procedures (with no clinically significant findings): physical exam, 12-lead ECG, or clinical laboratory tests
* Patient meets protocol criteria for diagnosis of IBS-C
* Patient demonstrates continued IBS-C through Pretreatment Period
* Patient is compliant with IVRS

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has symptoms of or been diagnosed with a medical condition that may contribute to abdominal pain
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Johnston, MD, FACP, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (100):
- United States (100):
  - Ironwood Investigational Site, Birmingham, Alabama
  - Ironwood Investigational Site, Huntsville, Alabama
  - Ironwood Investigational Site, Phoenix, Arizona
  - Ironwood Investigational Site, Tempe, Arizona
  - Ironwood Investigational Site, Tucson, Arizona
  - Ironwood Investigational Site, Sherwood, Arkansas
  - Ironwood Investigational Site, Anaheim, California
  - Ironwood Investigational Site, Chula Vista, California
  - Ironwood Investigational Site, Encinitas, California
  - Ironwood Investigational Site, Garden Grove, California
  - Ironwood Investigational Site, Laguna Hills, California
  - Ironwood Investigational Site, Orange, California
  - Ironwood Investigational Site, San Carlos, California
  - Ironwood Investigational Site, San Diego, California
  - Ironwood Investigational Site, Colorado Springs, Colorado
  - Ironwood Investigational Site, Bristol, Connecticut
  - Ironwood Investigational Site, Boynton Beach, Florida
  - Ironwood Investigational Site, Hollywood, Florida
  - Ironwood Investigational Site, Inverness, Florida
  - Ironwood Investigational Site, Jacksonville, Florida
  - Ironwood Investigational Site, Lauderdale Lakes, Florida
  - Ironwood Investigational Site, Miami, Florida
  - Ironwood Investigational Site, Pinellas Park, Florida
  - Ironwood Investigational Site, Tampa, Florida
  - Ironwood Investigational Site, Newnan, Georgia
  - Ironwood Investigational Site, Peoria, Illinois
  - Ironwood Investigational Site, Anderson, Indiana
  - Ironwood Investigational Site, Clive, Iowa
  - Ironwood Investigational Site, Davenport, Iowa
  - Ironwood Investigational Site, Mission, Kansas
  - Ironwood Investigational Site, Overland Park, Kansas
  - Ironwood Investigational Site, Topeka, Kansas
  - Ironwood Investigational Site, Baton Rouge, Louisiana
  - Ironwood Investigational Site, Metairie, Louisiana
  - Ironwood Investigational Site, Monroe, Louisiana
  - Ironwood Investigational Site, Shreveport, Louisiana
  - Ironwood Investigational Site, Annapolis, Maryland
  - Ironwood Investigational Site, Baltimore, Maryland
  - Ironwood Investigational Site, Hollywood, Maryland
  - Ironwood Investigational Site, Laurel, Maryland
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Traverse City, Michigan
  - Ironwood Investigational Site, Troy, Michigan
  - Ironwood Investigational Site, Plymouth, Minnesota
  - Ironwood Investigational Site, Jackson, Mississippi
  - Ironwood Investigational Site, Tupelo, Mississippi
  - Ironwood Investigational Site, Jefferson City, Missouri
  - Ironwood Investigational Site, Marlton, New Jersey
  - Ironwood Investigational Site, Albuquerque, New Mexico
  - Ironwood Investigational Site, Mineola, New York
  - Ironwood Investigational Site, Pittsford, New York
  - Ironwood Investigational Site, Asheboro, North Carolina
  - Ironwood Investigational Site, Asheville, North Carolina
  - Ironwood Investigational Site, Chapel Hill, North Carolina
  - Ironwood Investigational Site, Charlotte, North Carolina
  - Ironwood Investigational Site, Greensboro, North Carolina
  - Ironwood Investigational Site, Harrisburg, North Carolina
  - Ironwood Investigational Site, Hickory, North Carolina
  - Ironwood Investigational Site, Huntersville, North Carolina
  - Ironwood Investigational Site, New Bern, North Carolina
  - Ironwood Investigational Site, Statesville, North Carolina
  - Ironwood Investigational Site, Winston-Salem, North Carolina
  - Ironwood Investigational Site, Beachwood, Ohio
  - Ironwood Investigational Site, Cincinnati, Ohio
  - Ironwood Investigational Site, Dayton, Ohio
  - Ironwood Investigational Site, Mentor, Ohio
  - Ironwood Investigational Site, Sylvania, Ohio
  - Ironwood Investigational Site, Wadsworth, Ohio
  - Ironwood Investigational Site, Oklahoma City, Oklahoma
  - Ironwood Investigational Site, Yukon, Oklahoma
  - Ironwood Investigational Site, Lancaster, Pennsylvania
  - Ironwood Investigational Site, Levittown, Pennsylvania
  - Ironwood Investigational Site, Reading, Pennsylvania
  - Ironwood Investigational Site, Sellersville, Pennsylvania
  - Ironwood Investigational Site, Washington, Pennsylvania
  - Ironwood Investigational Site, Anderson, South Carolina
  - Ironwood Investigational Site, Charleston, South Carolina
  - Ironwood Investigational Site, Simpsonville, South Carolina
  - Ironwood Investigational Site, Summerville, South Carolina
  - Ironwood Investigational Site, Bristol, Tennessee
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Germantown, Tennessee
  - Ironwood Investigational Site, Kingsport, Tennessee
  - Ironwood Investigational Site, Nashville, Tennessee
  - Ironwood Investigational Site, Beaumont, Texas
  - Ironwood Investigational Site, El Paso, Texas
  - Ironwood Investigational Site, Fort Worth, Texas
  - Ironwood Investigational Site, Houston, Texas
  - Ironwood Investigational Site, Irving, Texas
  - Ironwood Investigational Site, Longview, Texas
  - Ironwood Investigational Site, San Antonio, Texas
  - Ironwood Investigational Site, Sugarland, Texas
  - Ironwood Investigational Site, Ogden, Utah
  - Ironwood Investigational Site, Salt Lake City, Utah
  - Ironwood Investigational Site, Chesapeake, Virginia
  - Ironwood Investigational Site, Lynchburg, Virginia
  - Ironwood Investigational Site, Spokane, Washington
  - Ironwood Investigational Site, Vancouver, Washington
  - Ironwood Investigational Site, La Crosse, Wisconsin
  - Ironwood Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Rao SS, Quigley EM, Shiff SJ, Lavins BJ, Kurtz CB, MacDougall JE, Currie MG, Johnston JM. Effect of linaclotide on severe abdominal symptoms in patients with irritable bowel syndrome with constipation. Clin Gastroenterol Hepatol. 2014 Apr;12(4):616-23. doi: 10.1016/j.cgh.2013.09.022. Epub 2013 Sep 25. PMID 24075889
- [Derived] Quigley EM, Tack J, Chey WD, Rao SS, Fortea J, Falques M, Diaz C, Shiff SJ, Currie MG, Johnston JM. Randomised clinical trials: linaclotide phase 3 studies in IBS-C - a prespecified further analysis based on European Medicines Agency-specified endpoints. Aliment Pharmacol Ther. 2013 Jan;37(1):49-61. doi: 10.1111/apt.12123. Epub 2012 Nov 1. PMID 23116208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over a fifteen month period from July 2009 to September 2010 at 111 US study sites.
Pre-assignment Details: Patients went through a 14 to 21 day Pretreatment Period during which the patients provided qualifying bowel habit and symptoms, and rescue medicine usage information through an interactive voice response system (IVRS). All randomized patients needed an abdominal pain score ≥ 3.
Groups:
- Placebo: Dose-matched placebo, oral administration, once per day.
- Linaclotide: Linaclotide 290μg, oral administration, once per day.
Period: Overall Study
Arm/Group | Placebo | Linaclotide
Started | 403 | 402
Completed | 305 | 294
Not Completed | 98 | 108
Not completed — Adverse Event | 10 | 41
Not completed — Protocol Violation | 11 | 8
Not completed — Withdrawal by Subject | 26 | 24
Not completed — Lost to Follow-up | 13 | 18
Not completed — Lack of Efficacy | 33 | 15
Not completed — Other reason | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide | Total
Number analyzed (Participants) | 403 | 402 | 805
Age Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.4) | 44.7 (13.1) | 44.3 (13.3)
Age, Customized [Number; unit: Participants]
  18 years 64 years | 386 | 379 | 765
  65 years and older | 17 | 23 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352 | 369 | 721
  Male | 51 | 33 | 84
Region of Enrollment [Number; unit: participants]
  United States | 403 | 402 | 805

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Pain and Complete Spontaneous Bowel Movement (APC) Responder, 9 Out of 12 Weeks
Description: A patient is considered to be a 9 out of 12 week APC responder if, for at least 9 out of the first 12 weeks of the treatment period, the patient had at least 3 CSBMs, had an increase of at least 1 CSBM from baseline, and had a decrease of at least 30 percent in their Abdominal Pain (AP) score from baseline during a particular week.
  The AP score assesses patient's worst AP in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no AP and 10 represents very severe AP.
  SBM is defined as a bowel movement that occurs in the absence of laxative, enema, or suppository use on either the calendar day of the bowel movement or the calendar day before the bowel movement. CSBM is defined as an SBM associated with a sense of complete evacuation.
Time Frame: Change from Baseline to Week 12
Population: 805 patients were randomized to treatment. 804 patients had at least 1 postrandomization entry of the primary efficacy assessment and were included in the Intent to Treat (ITT) Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
participants | 12 | 51
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 9/12 Week APC 3 + 1 Responders. The power, adjusted for multiplicity, was expected to be 93% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The p-value is still less than 0.05 after adjusting multiplicity using a serial gatekeeping multiple comparison procedure; Odds Ratio (OR) = 4.65, 95% CI 2-sided [2.44 to 8.84]

2. Primary Outcome: Complete Spontaneous Bowel Movement (CSBM) 3+1 Responder, 9 Out of 12 Weeks
Description: A patient is considered to be a CSBM 3+1 responder if, for at least 9 out of the 12 weeks of the treatment period, the patient had at least 3 CSBMs and experienced an increase of at least 1 CSBM from baseline during a particular week.
  A CSBM was defined as a Spontaneous Bowel Movement (SBM) that was associated with a sense of complete evacuation.
  An SBM was defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Change from Baseline to Week 12
Population: 805 patients were randomized to treatment. 804 patients had at least 1 postrandomization entry of the primary efficacy assessment and were included in the ITT Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
participants | 20 | 72
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 9/12 Week CSBM 3 + 1 Responders. The power, adjusted for multiplicity, was expected to be 93% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.19, 95% CI 2-sided [2.50 to 7.03]

3. Primary Outcome: Abdominal Pain Responder, 9 Out of 12 Weeks
Description: A patient is considered to be an abdominal pain responder if, for at least 9 out of the 12 weeks of the treatment period, they experienced a decrease of at least 30 percent in the mean abdominal pain score from baseline during a particular week.
  The Abdominal Pain score assesses patient's worst abdominal pain in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
participants | 79 | 156
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 9/12 Week Abdominal Pain Responders. The power, adjusted for multiplicity, was expected to be 93% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.91 to 3.60]

4. Primary Outcome: Abdominal Pain and Complete Spontaneous Bowel Movement (APC) Responder, 6 Out of 12 Weeks
Description: A patient is considered to be a 6 out of 12 week APC responder if, for at least 6 out of the first 12 weeks of the treatment period, the patient had an increase of at least 1 CSBM from baseline, and had a decrease of at least 30 percent in their Abdominal Pain (AP) score from baseline during a particular week.
  The AP score assesses patient's worst AP in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no AP and 10 represents very severe AP.
  SBM is defined as a bowel movement that occurs in the absence of laxative, enema, or suppository use on either the calendar day of the bowel movement or the calendar day before the bowel movement. CSBM is defined as an SBM associated with a sense of complete evacuation.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
participants | 56 | 135
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 6/12 Week APC + 1 Responders. The power, adjusted for multiplicity, was expected to be 86% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.16, 95% CI 2-sided [2.22 to 4.49]

5. Secondary Outcome: 12-Week Complete Spontaneous Bowel Movement (CSBM) Frequency
Description: The change from baseline in 12-week CSBM frequency (i.e., weekly CSBM frequency over the first 12 weeks of the Treatment Period).
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: CSBMs per Week
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
CSBMs per Week | 0.70 (0.12) | 2.24 (0.12)

6. Secondary Outcome: 12-Week Spontaneous Bowl Movement (SBM) Frequency
Description: The change from baseline in 12-week SBM frequency (i.e., weekly SBM frequency over the first 12 weeks of the Treatment Period).
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: SBMs per Week
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
SBMs per Week | 1.31 (0.18) | 4.02 (0.18)

7. Secondary Outcome: 12-Week Change in Stool Consistency
Description: The consistency of each BM was assessed by patients using the 7-point Bristol Stool Form Scale (BSFS) from 1 to 7.
  1. = separate hard lumps like nuts [difficult to pass]
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges [passed easily]
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces [entirely liquid]).
Time Frame: Change from Baseline to Week 12
Population: 805 patients were randomized to treatment; 804 patients had at least 1 postrandomization entry of the primary efficacy assessment and included in the ITT Population; 134 patients with no pretreatment spontaneous bowel movements were excluded from the Stool Consistency analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 332 | 338
Units on a scale | 0.61 (0.06) | 1.91 (0.06)

8. Secondary Outcome: 12-Week Change in Severity of Straining
Description: Straining is measured on a 5-point scale where a value of 1 is "not at all" and a value of 5 is "an extreme amount".
Time Frame: Change from Baseline to Week 12
Population: 805 patients were randomized to treatment; 804 patients had at least 1 postrandomization entry of the primary efficacy assessment and included in the ITT Population; 134 patients with no pretreatment spontaneous bowel movements were excluded from the Straining analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 332 | 338
Units on a scale | -0.66 (0.05) | -1.24 (0.04)

9. Secondary Outcome: 12-Week Change in Abdominal Pain Score
Description: Abdominal Pain at its worst (in the last 24 hours) is based on an 11-point scale where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
Units on a scale | -1.07 (0.09) | -1.85 (0.09)

10. Secondary Outcome: 12-Week Change in Abdominal Discomfort
Description: Abdominal discomfort was assessed on an 11-point scale where a value of 0 is "none" and a value of 10 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
Units on a scale | -1.10 (0.09) | -1.94 (0.09)

11. Secondary Outcome: 12-Week Change in Bloating
Description: Bloating was assessed on an 11-point scale where a value of 0 is "none" and a value of 10 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
Units on a scale | -1.03 (0.10) | -1.91 (0.09)

12. Secondary Outcome: Complete Spontaneous Bowl Movement (CSBM) Responder for 6 Weeks Out of 12 Weeks of Treatment
Description: A patient is considered to be a CSBM responder if, for at least 6 out of the 12 weeks of the treatment period, an increase of at least 1 CSBM per week from baseline was experienced.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
participants | 91 [2.29 to 4.21] | 191

13. Secondary Outcome: Abdominal Pain Responder for 6 Out of 12 Weeks
Description: A patient is considered to be an AP responder if, for at least 6 out of the first 12 weeks of the treatment period, the patient had a decrease of at least 30 percent in their Abdominal Pain score from baseline during a particular week.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
participants | 139 | 196

14. Secondary Outcome: 12-Week Percent of Abdominal Pain-free Days
Description: Abdominal pain free (APF) days are those days where the patient reported a score of '0' for abdominal pain at its worst.
  Abdominal Pain at its worst (in the last 24 hours) is based on an 11-point scale where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent of Pain-free Days
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 403 | 401
Percent of Pain-free Days | 4.83 (16.64) | 10.49 (23.42)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from July of 2009 to September of 2010 (26 weeks of safety data were collected)
Arm/Group | Placebo | Linaclotide
Serious Adverse Events (participants affected / at risk) | 7/403 | 4/402
Other Adverse Events (participants affected / at risk) | 86/403 | 137/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=403) | Linaclotide (N=402)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cystopexy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hodgkin's disease nodular sclerosis stage IVa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=403) | Linaclotide (N=402)
Diarrhea (Gastrointestinal disorders) | 10 | 79
Nausea (Gastrointestinal disorders) | 24 | 23
Sinusitis (Infections and infestations) | 28 | 23
Upper respiratory tract infection (Infections and infestations) | 22 | 22
Urinary tract infection (Infections and infestations) | 22 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that publication cannot be made for 24 months from the date of final data lock of the study, the sponsor can review the publication prior to public release, sponsor requires a minimum 60 day review period for each publication, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request an additional delay period of 60 days in order to protect potentially patentable information.